CLINICAL TRIAL: NCT05471869
Title: Computational Imaging Using Pixel-level Graph Adversarial Learning
Brief Title: Computational Imaging Research Based on Deep Learning
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xin Lou, professor, Chinese PLA General Hospital
Other Study IDs: Synthesis imaging-ChinaPLAGH
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Arterial Aneurysm
Keywords: Arterial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Aneurysm diagnosis — Intelligent detection and diagnosis of aneurysm diagnosis by CTA

SUMMARY:
Computational imaging research based on deep learning

DETAILED DESCRIPTION:
Based on the current technical challenges, subject development and upgrade of knowledge, to avoid the occurrence of adverse medical accidents, simplify the diagnostic process, artificial intelligence has become the alternative method of choice, by constructing training deep learning model, the CTA as model inputs aneurysm detection and diagnosis to improve diagnosis effectiveness, promote the development of medical technology

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-80 years.
2. CT paired imaging data of vessels, including layer-to-layer plain CT and enhanced CT. 2 Time range: January 2010 to December 2021.
3. Scanning sites: CT and CTA of head, neck, chest, abdomen or iliac.

Exclusion Criteria:

1. Unpaired CT image .
2. Severe artifact CT image.
3. enhancement CT failure image (failure to capture arterial phase or poor arterial development, insufficient flow of contrast agent, etc.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: varity of people
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-08-15 (Estimated)

PRIMARY OUTCOMES:
Objective evaluation | 30 minutes
  using SSIM\MAE index evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No